CLINICAL TRIAL: NCT05110469
Title: The Comparison of Intravenous Magnesium Sulphate and Intravenous Meperidine for Prevention of Shivering During Spinal Anesthesia
Brief Title: Comparison of MgSO4 Versus Meperidine for Prevention of Shivering During Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AnestesiaR (Other)
Responsible Party: Principal Investigator, Magdalena Sihombing, Principal Investigator, AnestesiaR
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MagnesiumAS01
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Shivering
Keywords: Magnesium sulphate; meperidine; shivering; spinal anesthesia
MeSH Terms: interventions — Magnesium Sulfate; Meperidine

STUDY DESIGN:
Intervention Model Description: Non-pregnant patients between 18-65 years of age, belonging to the American Society of Anesthesiologist physical status I or II who underwent spinal anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient allocation was done by randomization by anesthesiologists outside of the research team using randomization software. Patients would be divided into two groups, namely group M which contains MgSO4 30 mg/kg i.v. and group P which contains meperidine 0.5 mg/kg i.v. Anesthesiologists outside of the research team would prepare the study drug according to the randomized group. The formulated drug would be labeled as research drug without mentioning the content or group of the drug.
  Prior to spinal anesthesia, another OK team outside of the research team would give the research drug without knowing the contents of the drug, as well as perform spinal anesthesia. Observation of the data would be carried out by the researcher together with the OR team who performed the spinal anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Experimental): IV Magnesium sulphate 30 mg/kg in 100 ml NaCl 0.9%
  Interventions: Drug: Magnesium sulfate
- Group P (Experimental): IV Meperidine 0.5 mg/kg in 100 ml NaCl 0.9%
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: Magnesium sulfate — IV Magnesium sulphate 30 mg/kg, labeled as "research drug" for blinding, were given in 10 minutes while patients were monitored for side effects such as hypotension, bradycardia, nausea, vomiting, itch, allergy, drowsiness, and respiratory depression.
  Arms: Group M
Drug: Meperidine — IV Meperidine 0.5 mg/kg, labeled as "research drug" for blinding, were given in 10 minutes while patients were monitored for side effects such as hypotension, bradycardia, nausea, vomiting, itch, allergy, drowsiness, and respiratory depression.
  Arms: Group P

SUMMARY:
This was a double-blind randomized interventional study of 100 patients divided into two groups. Group M received MgSO4 30 mg/kg, and group P received meperidine 0.5 mg/kg intravenously in 100 ml of 0.9% NaCl before undergoing spinal anesthesia. Participants were non-pregnant patients between 18-65 years of age, belonging to the American Society of Anesthesiologist physical status I or II. Shivering was regarded as significant if it occurred at grade 3 or 4. Data of patient characteristics, shivering degree, tympanic membrane temperature, vital sign, and side effects were recorded.

DETAILED DESCRIPTION:
Study Design This was double-blinded randomized clinical trial that was conducted in Dr. Cipto Mangunkusumo National General Hospital in February - June 2021 after due permission from Ethics Committee of the Faculty of Medicine University of Indonesia - Cipto Mangunkusumo Hospital (No. KET-1510/UN2.F1/ETIK/PPM.00.02/2020). Patients were randomly devided into two groups to recieved MgSO4 30 mg/kg (group M) and meperidine 0.5 mg/kg (group P). Drugs will be prepared and delivered by another anesthesiologist outside of the research team.

Subjects Following patient informed consent, 100 patients aged 18-65 years old, with American Society of Anesthesiologist (ASA) physical status I or II who underwent spinal anesthesia. The following groups of patients were excluded from the study: patients with a history of allergy to the drugs used in the study, pregnant patients, neuromuscular disease, hyperthyroid, severe cardiopulmonary diseases, liver and/or renal disorders, used drugs that could interact with MgSO4 such as nifedipine, and preoperative body temperature less than 36oC or more than 37.5oC. Patients were dropped out if: any complications such as systemic allergic reaction, anaphylaxis, cardiac arrest was occured, failure of spinal anesthesia, respinal, surgery duration less than 30 minutes, and conversion to general anesthesia during evaluation.

Interventions and Outcomes After randomization, subjects would be given drugs according to their randomization group. MgSO4 30 mg/kg and meperidine 0.5 mg/kg were dissolved in 100 ml NaCl 0.9%, and labeled as "research drug" for blinding. Drugs were given in 10 minutes while patients were monitored for side effects such as hypotension, bradycardia, nausea, vomiting, itch, allergy, drowsiness, and respiratory depression. If hypotension occurs or blood pressure decreases >20% from baseline, patients will be treated with a crystalloid solution and intravenous ephedrine 5-10 mg.

Afterwards, patients were given 10 ml/kg crystalloid with room temperature 22oC - 23oC for 10 minutes before spinal anesthesia. Spinal anesthesia was performed at the lumbar vertebrae 3-4 or 4-5 interspaces, with 15 mg hyperbaric bupivacaine and fentanyl 25 mcg. Room temperature was maintained between 19oC - 24oC. Patients were covered with one layer of blanket, which covered the chest and upper arm, and other areas outside the operating area. Patients were given fluid maintenance of 2 ml/kg/hour crystalloid and oxygen supplementation 2-3 l/minute by nasal cannula. Patient ini this study also were managed in the state of Ramsay sedation scale 2 (co-operative, oriented, and tranquil) or 3 (appears asleep, but responds to verbal command), so some patient were given midazolam intravenously to maintain the condition.

The incidence of shivering, mean arterial pressure, heart rate, respiratory rate, and tympanic membrane temperature were observed every five minutes during the first 15 minutes and every 15 minutes within the next 120 minutes. The degree of shivering was measured with Crossley and Mahajan scale which is 0 = No shivering, 1 = piloerection or peripheral vasoconstriction, 2 = muscular activity in only 1 muscle group, 3 = muscular activity in more than 1 muscle group but not generalized, and 4 = intens shivering involving the whole body, except in the muscle affected by spinal block.6 Drugs were considered effective if they could prevent the incidence of 3rd or 4th degree shivering. Meperidine 25 mg intravenously was given if 3rd or 4th degree shivering occurred. Nausea and vomiting was treated by IV metoclopramide 10 mg. Postoperatively, all patients were transferred to recovery room and monitored for one hour until discharge.

Statistical Analysis All statistical analyses were performed using SPSS (Statistical Package for Social Sciences) version 20.0. Chi-square test or Fisher's exact test were used to compare the difference of proportion in shivering between the two groups. For numerical data, T-test and Mann-Whitney test were used. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old
* American Society of Anesthesiologist (ASA) physical status I or II
* Planning for spinal anesthesia

Exclusion Criteria:

* History of allergy to the drugs used in the study
* Pregnant patients
* With neuromuscular disease, hyperthyroid, severe cardiopulmonary diseases, liver and/or renal disorders
* Used drugs that could interact with MgSO4 such as nifedipine
* Preoperative body temperature less than 36oC or more than 37.5oC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Drug effectiveness | 120 minutes
  Drugs were considered effective if they could prevent the incidence of 3rd or 4th degree shivering

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo National General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No